CLINICAL TRIAL: NCT03588403
Title: Comparison of Tomotherapy Versus Intensity-modulated Radiotherapy for Patients With Nasopharyngeal Carcinoma: a Prospective,Phase II Study
Brief Title: TOMO Versus IMRT in Nasopharyngeal Carcinoma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiaozhong, chief phisician, Zhejiang Cancer Hospital
Other Study IDs: IRB-2018-133
Record Dates: First submitted 2018-07-04; First posted 2018-07-17 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A:Tomotherapy: Patients with non-disseminated nasopharyngeal carcinoma receiving Tomotherapy.The prescribed radiation dose was defined as follows: PGTVnx 7040cGy/32F,PGTVnd 7040cGy/32F,PTV1 6080cGy/32F,PTV2 5440cGy/32F.
  Interventions: Radiation: TOMO
- Arm B: IMRT: Patients with non-disseminated nasopharyngeal carcinoma receiving IMRT.The prescribed radiation dose was defined as follows: PGTVnx 7040cGy/32F,PGTVnd 7040cGy/32F,PTV1 6080cGy/32F,PTV2 5440cGy/32F.
  Interventions: Radiation: IMRT

INTERVENTIONS:
Radiation: TOMO — Tomotherapy
  Groups: Arm A:Tomotherapy
Radiation: IMRT — Intensity modulated radiotherapy
  Groups: Arm B: IMRT

SUMMARY:
Tomotherapy is a new radiation planning and delivery technology which may allow for delivery of higher radiation doses with less damage to normal tissues. The investigators aim to compare the treatment efficacy and quality of life between tomotherapy and intensity-modulated radiotherapy for patients with nasopharyngeal carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed non-keratinizing carcinoma.
2. Tumor staged T1-4N0-3M0 （according to the 8th AJCC staging system）
3. Performance status: KPS>70
4. With normal liver function test (ALT, AST <1.5ULN)
5. Renal: creatinine clearance >60ml/min
6. Without hematopathy,marrow: WBC >4*109/L, HGB>80G/L, and PLT>100*109/L.
7. Written informed consent

Exclusion Criteria:

1. WHO type I squamous cell carcinoma or adenocarcinoma
2. Age >65 or <18
3. Prior malignancy (except adequately treated carcinoma in-situ of the cervix or basal/squamous cell carcinoma of the skin)
4. Previous chemotherapy or radiotherapy (except non-melanomatous skin cancers outside the intended RT treatment volume)
5. Patient is pregnant or lactating
6. Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), and emotional disturbance.

   -

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: nasopharyngeal carcinoma patients staged T1-4N0-3M0
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
QoL(quality of life) | 2 years
  Changes in quality of life were assessed by EORTC QLQ-C30

SECONDARY OUTCOMES:
PFS (progression free survival) | 2 years
  from the first day of therapy to the date of disease progression or death from any cause, whichever was first (according the criterion of RECIST 1.1 ).
OS (overall survival) | 2 years
  from the first day of therapy to death or last follow-up
LRRFS(Locoregional failure-free survival) | 2 years
  from the first day of therapy to the date of first locoregional relapse or until the date of the last follow-up visit.
Adverse Events | 5 years
  Participants will be followed for the duration of hospital stay, an expected average of 50 days and every 3 months thereafter for 5 years. Observe and record the toxicity profile (including but not limit to mucositis, liver and kidney function, et al.) according NCI-CTCAE 4.03 during the chemoradiation and follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaozhong Chen, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided